CLINICAL TRIAL: NCT04326426
Title: ODYSSEY: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy of Tradipitant in Treating Inflammatory Lung Injury and Improving Clinical Outcomes Associated With Severe or Critical COVID-19 Infection
Brief Title: ODYSSEY: A Study to Investigate the Efficacy of Tradipitant in Treating Severe or Critical COVID-19 Infection
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLY-686-3501
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tradipitant (Experimental): Tradipitant 85 mg PO BID
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): 2 capsules of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Neurokinin-1 antagonist
  Arms: Tradipitant
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind placebo-controlled trial to investigate the efficacy and safety of tradipitant 85 mg orally given twice daily to treat inflammatory lung injury associated with severe or critical COVID-19 infection.

On evaluation for enrollment, participant will need to meet all inclusion and exclusion criteria. If participant consents, they will be randomized 1:1 to treatment with either tradipitant 85 mg PO BID or placebo in addition to standard of care for COVID-19 infection as per the protocol at the treating hospital. NEWS 2 will be assessed at screening and daily following randomization. Inflammatory lab markers as detailed should be collected once per day in the morning, preferably at the same time every morning. All enrolled participants will have whole blood collected for whole genome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-90
* Confirmed laboratory COVID-19 infection by RT-PCR
* Meeting severe or critical criteria of COVID-19 infection as defined at treating hospital
* Confirmed pneumonia by chest radiograph or computed tomography
* Fever defined as temperature ≥ 36.6 °C armpit, ≥ 37.2 °C oral, or ≥ 37.8 °C rectal
* Oxygen saturation less than 92%

Exclusion Criteria:

* Recent use of illicit drugs or alcohol abuse
* Known allergy to tradipitant or other neurokinin-1 antagonists
* Pregnancy
* Known HIV, HBV, or HCV infection
* Malignant tumor, other serious systemic diseases
* Inability to provide informed consent or to have an authorized relative or designated person provide informed consent, or to comply with the protocol requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to improvement on a 7-point ordinal scale as compared to baseline | 14 days or discharge

SECONDARY OUTCOMES:
Treatment and prevention of inflammatory lung injury as measured by change in baseline of interleukin-6 (IL-6) | 14 days or discharge
Rate of Decline of COVID-19 viral load assessed by RT-PCR from nasopharyngeal samples | 14 days or discharge
In-hospital mortality | 14 days or discharge
Mean change in NEWS2 score from baseline | 14 days or discharge
Understand the effect of genetics for treatment response through whole genome sequence of the participant and the COVID-19 virus | 14 days or discharge
Reduction from baseline of NRS for cough | 14 days or discharge
Reduction from baseline of NRS for nausea | 14 days or discharge
Time to normalization of fever for at least 48 hours | 14 days or discharge
Time to improvement in oxygenation for at least 48 hours | 14 days or discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Hospital Northwell Health, New York, New York, United States

REFERENCES:
- [Derived] Smieszek SP, Przychodzen BP, Polymeropoulos VM, Polymeropoulos CM, Polymeropoulos MH. Assessing the potential correlation of polymorphisms in the IL6R with relative IL6 elevation in severely ill COVID-19 patients'. Cytokine. 2021 Dec;148:155662. doi: 10.1016/j.cyto.2021.155662. Epub 2021 Jul 29. PMID 34353696